CLINICAL TRIAL: NCT05890417
Title: Evolution of Sexual Life Quality of Women With POI Before and After Introduction of Hormone Replacement Therapy
Acronym: SEX-POInt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2023/04
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Premature Ovarian Failure
Keywords: premature ovarian insufficiency; sexuality; quality of life
MeSH Terms: conditions — Primary Ovarian Insufficiency; Sexuality | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaires (Experimental): Female Sexual Function Index (FSFI) and WHO Quality of Life-BREF (WHOQOL-BREF) questionnaires at baseline and at 6 months after starting hormone replacement therapy.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Female Sexual Function Index (FSFI) and WHO Quality of Life-BREF (WHOQOL-BREF) questionnaires at baseline and 6 months after starting hormone replacement therapy

SUMMARY:
The aim of this study is to evaluate the evolution of quality of sex life of women with POI after introduction hormone replacement therapy through the FSFI scale

DETAILED DESCRIPTION:
Premature ovarian failure (POI) is a pathology that affects about 1-2% of women before the age of 40. The resulting estrogen deficiency is the cause of multiple repercussions. Clinically, sexual disorders may appear in the short term, such as a decrease in libido, vaginal dryness, an increase in dyspareunia, resulting in less frequent sexual intercourse and less satisfaction with sexual life. The quality of life of these patients also appears to be reduced compared to women with normal ovarian reserve. A 2008 study showed that the sexual function of patients with POI treated with hormone replacement therapy (HRT) was normal but remained significantly lower than that of patients with normal ovarian function. However, no study has attempted to assess the evolution of the symptomatology of these patients before and after the introduction of HRT. Evidence of improvement in sexual disorders under treatment could be an additional argument to improve patient adherence and treatment compliance; as well as information for health professionals

ELIGIBILITY:
Inclusion Criteria:

* positive diagnosis of POI (amenorrhea > 4 months or spaniomenorrhea > 4 months and FSH > 25 IU/L checked twice, more than 4 weeks apart)
* absence of hormonal treatment,
* patient's oral consent,
* affiliated or beneficiary of health insurance

Exclusion Criteria:

* contraindication to hormonal treatment (history of hormone-dependent cancer, history of ischemic arterial stroke),
* inability of the patient to understand the nature or risks or significance and implications of the clinical investigation,
* patient under legal protection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
FSFI questionnaire score | Month 6
  This is a self-assessment questionnaire with 19 items. It considers 6 domains of female sexuality: desire (2 items), arousal (4 items), lubrication (4 items), orgasm (3 items), satisfaction (3 items) and pain (3 items). The items are rated on a 0 or 1 to 5 point scale (low score of 0-1 to high score of 5) to determine a raw score per domain. Then, the score for each domain is multiplied by a standardised coefficient to arrive at a total score between 2 and 36.
  The cut-off point for differentiating between women with and without sexual problems is 26.55; a lower score reflects the existence of sexual problems.

SECONDARY OUTCOMES:
FSFI score according to the aetiology and to the mode of administration of hormonal treatment | Baseline, Month 6
  FSFI score before and after 6 months of treatment according to the aetiology of Premature ovarian failure (POI) (idiopathic, genetic, iatrogenic, Turner syndrome) and according to the mode of administration of hormonal treatment
WHOQOL-BREF score | Baseline, Month 6
  The WHOQOL-BREF questionnaire is a self-assessment questionnaire with 26 items and has been used to study the quality of life of patients with POI.
  The WHOQOL-BREF is the short version of the WHOQOL and addresses 4 domains of quality of life: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall quality of life and general health.
  The items are evaluated on a 5-point Likert scale (low score of 1 to high score of 5) to determine a raw score per item. Next, the average score for each domain is calculated, resulting in an average domain score between 4 and 20. Finally, this average domain score is then multiplied by 4 to transform the domain score into a scaled score (comparable to the score used in the original WHOQOL-100), with a higher score indicating a better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No